CLINICAL TRIAL: NCT00958399
Title: Satiety, Glycemic, and Gastrointestinal Effects of Novel Fibers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Tate and Lyle Ingredients France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 0701M00264
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: satiety; fiber; food intake; gut hormones; visual analog scales; microflora
MeSH Terms: interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- No fiber (Placebo Comparator): No fiber added to study products
  Interventions: Dietary Supplement: Placebo
- Resistant Starch (Experimental): Muffins, cereal, and bars made with a resistant starch
  Interventions: Dietary Supplement: Resistant Starch
- Resistant starch + soluble fiber (Experimental): Muffins, cereal, and bars made with a mixture of resistant starch and a soluble fiber
  Interventions: Dietary Supplement: Resistant starch + soluble fiber
- Fiber made from corn starch (Experimental): Muffins, cereal, and bars made with novel corn fiber
  Interventions: Dietary Supplement: Fiber made from corn starch
- Fiber made from corn starch + soluble fiber (Experimental): Muffins, cereal, and bars made with a mixture of novel corn fiber and a soluble fiber
  Interventions: Dietary Supplement: Fiber made from corn starch + soluble fiber

INTERVENTIONS:
Dietary Supplement: Placebo — Low fiber muffin, hot cereal and beverage (acute phase) or fiber bars and beverage (chronic phase)
  Arms: No fiber
Dietary Supplement: Resistant Starch — 25 g resistant starch, administered in a muffin, hot cereal and beverage (acute phase) or fiber bars and beverage (chronic phase)
  Arms: Resistant Starch
Dietary Supplement: Resistant starch + soluble fiber — 25 g fiber as resistant starch and a soluble fiber, administered in a muffin, hot cereal and beverage (acute phase) or fiber bars and beverage (chronic phase)
  Arms: Resistant starch + soluble fiber
Dietary Supplement: Fiber made from corn starch — 25 g fiber made from corn starch, administered in a muffin, hot cereal and beverage (acute phase) or fiber bars and beverage (chronic phase)
  Arms: Fiber made from corn starch
Dietary Supplement: Fiber made from corn starch + soluble fiber — 25 g fiber as a fiber made from corn starch and a soluble fiber, administered in a muffin, hot cereal and beverage (acute phase) or fiber bars and beverage (chronic phase)
  Arms: Fiber made from corn starch + soluble fiber

SUMMARY:
Research suggests dietary fiber may play a role in weight management, and fiber consumption is inversely associated with body weight, body fat, and BMI in cross-sectional studies. These effects may be mediated by increased satiety, reduced food intake, or changes in blood levels of glucose, insulin, and gut hormones.

The purpose of this study is to determine the satiety, glycemic, hormonal, and gastrointestinal responses of novel fiber supplements.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age 18-60 years
* non-smoking
* not taking medication
* non-dieting (weight stable in prior 3 months)
* BMI 18-27
* English literacy
* ability to give blood

Exclusion Criteria:

* do not regularly consume breakfast
* food allergies to ingredients found in study products
* dislike for muffins, fiber bars, or hot cereal
* BMI <18 or >27
* diagnosed cardiovascular, renal, or hepatic disease
* diabetes mellitus (fasting blood sugar >126 mg/dl)
* cancer in previous 5 years (except basal cell carcinoma of the skin)
* any gastrointestinal disease or condition
* recent bacterial infection (< 3 months)
* recent or concurrent participation in an intervention research study
* history of drug or alcohol abuse in prior 6 months
* use of lipid-lowering, anti-hypertensive, or anti-inflammatory steroid medication
* restrained eaters
* vegetarians
* people who eat more than approximately 15 grams of fiber per day
* women who are pregnant or lactating
* women with irregular menstrual cycles

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Satiety | 0, 15, 30, 45, 60, 90, 120, 180, 215 minutes postprandially

SECONDARY OUTCOMES:
ad libitum food intake | 180 minutes postprandially and over 24 hours
Ghrelin, polypeptide YY (PYY), and glucagon-like peptide-1 (GLP-1) response | 0, 30, 60 minutes postprandially
Gastrointestinal tolerance and fecal chemistry | following 7 days of treatment
Glucose/Insulin Response | 0, 15, 30, 45, 60, 90, 120, 180 minutes postprandially

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota - General Clinical Research Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Timm DA, Thomas W, Boileau TW, Williamson-Hughes PS, Slavin JL. Polydextrose and soluble corn fiber increase five-day fecal wet weight in healthy men and women. J Nutr. 2013 Apr;143(4):473-8. doi: 10.3945/jn.112.170118. Epub 2013 Feb 20. PMID 23427334